CLINICAL TRIAL: NCT07128654
Title: A Randomized, Open, Single-dose, Crossover-design, Phase I Study to Evaluate the Safety and Pharmacokinetics After Co-administration of CTL0201 and CTL0202 or Administration of CT-L02 in Healthy Volunteers
Brief Title: A Bioequivalence Study of CT-L02 Compared to Co-administration (CTL0201 and CTL0202) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT-L02-102
Record Dates: First submitted 2025-08-14; First posted 2025-08-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): CTL02
  Interventions: Drug: CTL02
- Arm B (Active Comparator): Co-administration of CTL0201 and CTL0202
  Interventions: Drug: CTL0201; Drug: CTL0202

INTERVENTIONS:
Drug: CTL02 — FDC tablet, single dose, oral administration
  Arms: Arm A
Drug: CTL0201 — Nesina, tablet, single dose, oral administration
  Arms: Arm B
Drug: CTL0202 — Jardiance, tablet, single dose, oral administration
  Arms: Arm B

SUMMARY:
This is a randomized, open, single-dose, crossover-design, phase I study to evaluate the safety and pharmacokinetics after co-administration of CTL0201 and CTL0202 or administration of CT-L02 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant aged 19 to 55 years, at screening
* A participant who has a body mass index (BMI) of 18.0~29.9 kg/m2, at screening
* A participant who is judged to be eligible to participate by the results of screening tests (vital signs, clinical laboratory tests, 12-lead ECG, etc.) by the principal investigator

Exclusion Criteria:

* A participant who has taken drugs that induce or inhibit drug metabolizing enzymes
* A participant who has participated in other clinical trials or bioequivalence studies within 6 months prior to the first dose of the investigational drug
* A participant who has a history of gastrointestinal surgery that may affect drug absorption

Ages: 19 Days to 55 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-10-26 (Actual)

PRIMARY OUTCOMES:
AUCt (Area under the plasma concentration-time curve) | 0(Pre-dose), 0.17, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 48, 72hrs
Cmax (Peak Plasma Concentration) | 0(Pre-dose), 0.17, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 48, 72hrs

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, South Korea